CLINICAL TRIAL: NCT06248996
Title: ARTSCAN VI Protocol Version 1, 2023-07-03 ARTSCAN VI - a Multicentre Phase III Study of Risk-based Treatment Intensification With Hyperfractionated Radiotherapy in Head and Neck Cancer Patients
Brief Title: a Multicentre Phase III Study of Risk-based Treatment Intensification With Hyperfractionated Radiotherapy in Head and Neck Cancer Patients
Acronym: ARTSCAN VI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARTSCAN VI
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Head and neck squamous cell carcinoma; radiotherapy; HNSCC; Hyperfractionated radiotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventionally fractioned (standard) group (Active Comparator): This groups is treated with standard radiotherapy treatment: RT 2.0 Gy daily to final radiation dose 68.0 Gy or
  Interventions: Radiation: Control group
- HFX-RT group (Experimental): Treated with Hyperfractionated radiotherapy (HFX-RT): Gy twice daily (10 fractions/week) with final dose 83.0 Gy
  Interventions: Radiation: Hyperfractionated radiotherpy

INTERVENTIONS:
Radiation: Hyperfractionated radiotherpy — 83.0 Gy in 68 fractions, 1.22 Gy per fraction, two daily fractions, five days per week to the primary tumour volume (GTVT_83.0). To the primary tumour with an added margin (PTVT_74.8) and to neck node metastases (PTVN_74.8) the prescribed dose will be 74.8 Gy in 68 fractions, 1.10 Gy per fraction twice daily. To elective neck nodes (PTV 54.4) the prescribed dose will be 54.4 Gy in 68 fractions, 0.80 Gy per fraction twice daily.
  Other Names: HFX-RT
  Arms: HFX-RT group
Radiation: Control group — 68.0 Gy in 34 fractions, 2.00 Gy per fraction per day, five or six days per week to tumour volumes and 54.4 Gy in 34 fractions, 1.60 Gy per fraction to elective neck nodes.
  Other Names: standard treatment
  Arms: Conventionally fractioned (standard) group

SUMMARY:
There is an unmet need to personalise treatment for patients with head and neck squamous cell carcinoma (HNSCC) and to improve treatment results for patients with advanced disease. In this phase III study, HNSCC patients with prognostic factors indicating increased risk of treatment failure that are aimed for curative treatment with radiotherapy (RT) will be randomised between standard treatment (conventionally fractionated RT with final RT dose 68.0 Gy) and hyperfractionated RT (HFX-RT) with final RT dose 83.0 Gy.

In order to find better prognostic and predictive tools the study also includes exploratory and translational analyses including evaluation of grade of hypoxia with Magnetic Resonance Imaging (MRI) and gene profiling by RNA-sequencing, tumour immune profiling, comparisons of global gene expression, gene aberrations and protein expression, and texture analyses of CT, FDG-PET and MRI images used during RT preparation and during patient follow-up. Patients with tumours with lower risk of recurrence, not eligible for randomisation in the study, can still participate in the translational parts of the study not investigating response to altered fractionation.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be at least 18 years old.
2. Histologically or cytologically confirmed, previously untreated, HNSCC of the oropharynx, hypopharynx, larynx or oral cavity without distant metastases and aimed for treatment with radiotherapy (with or without concomitant chemotherapy) with curative intent.
3. The primary tumour must fulfil the following high-risk criteria:

   1. For p16+ oropharyngeal cancer: Radiographic measurement of threeorthogonal diameters must render a tumour estimate of ≥30 cc.
   2. For all other subsites and for p16- oropharyngeal cancer: Radiographic measurement of three orthogonal diameters must render a tumour estimate of ≥20 cc.
4. The treatment may be followed but not preceded by surgery, either as a salvage procedure or a neck dissection. An excision of a lymph node or tonsillectomy for diagnostic purposes, does not exclude the patient from participation.
5. WHO/ECOG performance status 0-2
6. The patient must be able to understand the information about the treatment and give a written informed consent to participate in the trial.

Exclusion Criteria:

1. Previous radiotherapy in the head and neck region.
2. Concomitant or previous malignancies, except uncomplicated basal cell carcinoma, early (T1-2 N0) squamous cell carcinoma of the skin with follow-up time of at least one year for squamous cell carcinomas, and except other cancer with a disease-free follow-up of at least three years
3. Two or more synchronous primary HNSCC at time of diagnosis
4. Nasopharyngeal cancer
5. Sinonasal cancer
6. Co-existing disease prejudicing survival (expected survival < three years).
7. Pregnancy or lactation
8. Psychiatric or addictive disorders or other medical conditions which in the view of the investigator might impair patient compliance

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2028-03-04 (Estimated); Study Completion 2033-03-04 (Estimated)

PRIMARY OUTCOMES:
Local tumour control after treatment | Every three months for two years, then every 6 moths up to 5 years
  Local tumour control after treatment with conventionally fractionated (standard) RT compared with hyperfractionated radiotherapy (HFX-RT)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Gebre-Medhin, MD, Principal Investigator — Lund University Hospital
Locations (11):
- Sweden (11):
  - Gävle Hospital, Gävle
  - Sahlgrenska University Hospital, Gothenburg
  - Jönköping Hospital, Jönköping
  - Karlstad Hospital, Karlstad
  - Linköping University hospital, Linköping
  - Lund University Hospital, Lund
  - Örebro University Hospital, Örebro
  - Karolinska University Hospital, Stockholm
  - University Hospital, Umeå
  - Uppsala Accademical Hospital, Uppsala
  - Västmanlands Hospital Västerås, Västerås